CLINICAL TRIAL: NCT00082082
Title: A Trial of Thymalfasin With Trans Arterial Chemo-Embolization (TACE) in the Treatment of Adult Patients With Unresectable Hepatocellular Carcinoma: A Phase II Trial
Brief Title: A Trial of Thymalfasin in Adult Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SciClone Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ta1-HCC-2K1001
Record Dates: First submitted 2004-04-28; First posted 2004-04-30 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Thymalfasin

INTERVENTIONS:
Drug: Thymalfasin (thymosin alpha-1)
Procedure: Trans arterial chemoembolization (TACE)

SUMMARY:
The objective of this Phase II trial is to compare the efficacy and safety of 6 months of treatment with thymalfasin plus trans arterial chemoembolization (TACE) with TACE alone in adult patients with non-surgical hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Diagnosis of HCC by:

  1. Presence of HCC on biopsy (core biopsy), or, if biopsy is strongly contra-indicated due to safety or patient-related concerns, then the diagnosis of HCC can be determined by:
  2. A new hepatic defect on imaging with an AFP > 1000 ng/ml, or
  3. A new hepatic defect on ultrasound or CT with an AFP < 1000 ng/ml when one of the following is present:

     1. At least two additional imaging techniques show signs characteristic of HCC, or
     2. The new hepatic defect has doubled in diameter over time, or
     3. The AFP has progressively risen to > 200 ng/ml and triples the mean baseline.
* HCC must be unresectable and non-transplantable.
* Hematocrit > 30%, platelet count >= 50,000 per microliter, WBC > 2.0 x 109/L, and polymorphonuclear white cell count >= 1.0 x 109/L.
* Adequate renal function as demonstrated by serum creatinine level < 1.5 mg/dl.
* If the patient is a woman, she is using a definitive method of birth control in consultation with her physician, or is surgically sterile or post-menopausal.

Exclusion Criteria:

* Concomitant chronic use of any drug known to be hepatotoxic, or of any immunosuppressive drug (Use of oral contraceptives will not exclude an otherwise eligible patient).
* Presence of main portal vein thrombosis or hepatic artery malformation.
* HCC amenable to treatment by surgical resection or hepatic transplantation.
* HIV infection diagnosed by HIV seropositivity and confirmed by Western blot.
* Concomitant or prior history of malignancy other than HCC within the last 10 years, except for curatively treated skin cancer or surgically cured in situ carcinoma of the cervix.
* Active infectious process that is not of a self-limiting nature. TB and AIDS are examples of infectious processes that are not of a self-limiting nature.
* Pregnancy as documented by a urine pregnancy test. Women with reproductive potential must agree to practice an adequate method of birth control for the duration of the study.
* Alcohol or intravenous drug abuse within the previous 1 year.
* Previous treatment with thymalfasin.
* Patients with known hypersensitivity to iodine.
* Simultaneous participation in another investigational drug study, or participation in any clinical trial involving investigational drugs within 30 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - California Pacific Medical Center, San Francisco, California
  - University of Florida, Gainesville, Florida
  - William Beaumont Hospital, Royal Oak, Michigan
  - Columbia University, New York, New York
  - Metropolitan Research, Fairfax, Virginia